CLINICAL TRIAL: NCT03631719
Title: World Mosquito Program - Colombia (WMP-COLOMBIA): The Impact of City-wide Deployment of Wolbachia-infected Mosquitoes on Arboviral Disease Incidence in Medellin and Bello, Colombia
Brief Title: Impact of Wolbachia Deployment on Arboviral Disease Incidence in Medellin and Bello, Colombia
Acronym: WMP-COL
Status: Completed | Type: Observational
Sponsor: Universidad de Antioquia (Other)
Collaborators: Monash University (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PEC004_18; PECET-002 (Registry Identifier: Impact Assessment of Wolbachia deployment)
Record Dates: First submitted 2018-07-13; First posted 2018-08-15 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Chikungunya Virus Infection; Zika Virus Infection
Keywords: Wolbachia; Colombia; Dengue; Zika; Chikungunya; Arboviral diseases; Disease surveillance
MeSH Terms: conditions — Dengue; Chikungunya Fever; Zika Virus Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — 6 ml venous blood sample for DENV, chikungunya virus (CHIKV), and Zika virus (ZIKV) diagnostic testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early-release: Resident in areas that receive early Wolbachia deployments.
  Interventions: Biological: Wolbachia-carrying Ae.aegypti mosquitoes
- Late-release: Resident in areas that receive late Wolbachia deployments.

INTERVENTIONS:
Biological: Wolbachia-carrying Ae.aegypti mosquitoes — Wolbachia-infected Ae. aegypti mosquito eggs and adults sequentially deployed into Medellin and Bello, Colombia. Deployments cease once Wolbachia prevalence has reached a predetermined frequency (usually ≥60%).
  Groups: Early-release

SUMMARY:
Study setting: Medellin and Bello municipalities, Colombia Health condition(s) studied: Dengue, Zika and chikungunya virus infection Intervention: Deployment of Wolbachia-infected Aedes aegypti mosquitoes in Medellin and Bello.

Study design:

1. An interrupted time-series analysis utilising routine disease surveillance data collected by the Medellín and Bello Health Secretariats, which aims to compare incidence of dengue, chikungunya and Zika pre- and post-Wolbachia release.
2. A test-negative study using an incident case-control design, which aims to quantify the reduction in disease incidence among people living within a Wolbachia-treated zone compared with an untreated zone that has a similar dengue risk profile at baseline.

DETAILED DESCRIPTION:
* Selection and enrolment of participants: Enrolment of patients will commence after completion of Wolbachia releases in the early zones. Study processes for enrolling patients presenting with febrile illness will be established at a network of primary health care facilities that serve the population who reside in the study area. Trained research staff will be employed to assist with study processes in each site. Participants will be enrolled from within the population of patients (aged ≥3 years old) presenting with undifferentiated fever of 1-4 days' duration. All patients meeting the inclusion criteria will be eligible for enrolment and will be asked to provide written informed consent before participating in the study.
* Recruitment procedures: All eligible participants meeting study inclusion criteria will be invited to enroll continuously throughout the study period. Recruitment will occur during normal clinic hours. Participants will be managed according to standard clinical practice by the attending physicians. Recruitment rates in each clinic and across the study site as a whole will be monitored weekly, including a review of the screening logs to identify the proportion of eligible participants who did not consent to participate. The field coordinator will make regular visits to low-enrolling clinics to identify clinic-based, patient-based or other causes for low recruitment, and put measures in place to address these.
* Screening: All patients presenting with febrile illness will be screened against the study inclusion criteria by trained staff. All eligible febrile individuals will be recorded in a screening log and invited to participate. Participation status (consent/decline) will be recorded against each participant in the log.
* Informed consent: Written informed consent will be sought from participants (or their guardian where the participant is a minor) by trained local staff, after explaining the study objectives, processes, data, and sample collection, and the participant has had an opportunity to ask questions. A verbal explanation of the written Explanatory Statement will be provided to all participants in the local language. In addition, participants aged between 7 and 17 years will be invited to sign an assent form indicating they understand the research and agree to participate. Data and sample collection procedures
* Data collection: A unique identifier will be assigned to each participant at enrollment. Basic demographic details, eligibility against the inclusion criteria and illness onset date will be recorded in a standardized case report form.

ELIGIBILITY:
Inclusion Criteria:

* Fever (either self-reported or objectively measured, e.g. axillary temperature ≥38oC, with a date of onset between 1-4 days prior to the day of presentation.
* Aged ≥3 years old.
* Lived (i.e. slept) in the study area every night (or day) for the 10 days preceding illness onset.

Exclusion Criteria:

* Localising features suggestive of a specific diagnosis e.g. severe diarrhea, otitis, pneumonia
* Prior enrollment in the study within the previous 4 weeks.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The case-control study area as a whole has a population of approximately 564,000, of which approximately half will be resident in areas that receive early Wolbachia deployments ('early-release') and half in areas that will receive late Wolbachia deployments ('late-release').
  The study population for measurement of the efficacy endpoint is the population of patients who reside in the study area, presenting to the network of participating primary health care facility with febrile illness, and meeting the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 834 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Dengue cases notified to surveillance system | 5 years
  Incidence of dengue cases (suspected, epidemiological link, and IgM positive for dengue) notified to the disease surveillance system
Virologically-confirmed dengue | 2 years
  Virologically-confirmed dengue virus infection in patients reporting febrile illness recruited from health clinics. Participants are classified as dengue cases if plasma samples collected 1-4 days after onset of fever test positive for dengue virus NS1 antigen or dengue virus nucleic acid by RT-qPCR.

SECONDARY OUTCOMES:
IgM test positive for dengue | 5 years
  Number of cases who were IgM test positive for dengue
Severe dengue cases | 5 years
  Incidence of severe dengue cases reported to the surveillance system, by release zone and overall.
Zika cases notified to surveillance system | 5 years
  Incidence of Zika cases reported to the surveillance system.
Chikungunya cases notified to surveillance system | 5 years
  Incidence of chikungunya cases reported to the surveillance system.
Spatial analysis | 5 years
  The spatial distribution of notified dengue cases with geolocated primary address available, before and after Wolbachia deployment
Virologically-confirmed chikungunya infection | 2 years
  Virologically-confirmed chikungunya virus infection in patients reporting febrile illness recruited from health clinics. Participants are classified as chikungunya cases if plasma samples collected 1-4 days after onset of fever test positive for chikungunya virus NS1 antigen or chikungunya virus nucleic acid by RT-qPCR.
Virologically-confirmed Zika infection | 2 years
  Virologically-confirmed Zika virus infection in patients reporting febrile illness recruited from health clinics. Participants are classified as Zika cases if plasma samples collected 1-4 days after onset of fever test positive for Zika virus NS1 antigen or Zika virus nucleic acid by RT-qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Simmons, Prof., Study Director — Monash University
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brady OJ, Gething PW, Bhatt S, Messina JP, Brownstein JS, Hoen AG, Moyes CL, Farlow AW, Scott TW, Hay SI. Refining the global spatial limits of dengue virus transmission by evidence-based consensus. PLoS Negl Trop Dis. 2012;6(8):e1760. doi: 10.1371/journal.pntd.0001760. Epub 2012 Aug 7. PMID 22880140
- [Background] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Background] Shepard DS, Coudeville L, Halasa YA, Zambrano B, Dayan GH. Economic impact of dengue illness in the Americas. Am J Trop Med Hyg. 2011 Feb;84(2):200-7. doi: 10.4269/ajtmh.2011.10-0503. PMID 21292885
- [Background] Shepard DS, Undurraga EA, Halasa YA. Economic and disease burden of dengue in Southeast Asia. PLoS Negl Trop Dis. 2013;7(2):e2055. doi: 10.1371/journal.pntd.0002055. Epub 2013 Feb 21. PMID 23437406
- [Background] Shepard DS, Suaya JA, Halstead SB, Nathan MB, Gubler DJ, Mahoney RT, Wang DN, Meltzer MI. Cost-effectiveness of a pediatric dengue vaccine. Vaccine. 2004 Mar 12;22(9-10):1275-80. doi: 10.1016/j.vaccine.2003.09.019. PMID 15003657
- [Background] Dengue Vaccine Initiative. Dengue vaccine candidates in clinical development. (2016). Available at: http://www.denguevaccines.org/vaccine-development. (Accessed: 13th June 2016)
- [Background] L'Azou M, Moureau A, Sarti E, Nealon J, Zambrano B, Wartel TA, Villar L, Capeding MR, Ochiai RL; CYD14 Primary Study Group; CYD15 Primary Study Group. Symptomatic Dengue in Children in 10 Asian and Latin American Countries. N Engl J Med. 2016 Mar 24;374(12):1155-66. doi: 10.1056/NEJMoa1503877. PMID 27007959
- [Background] Capeding MR, Tran NH, Hadinegoro SR, Ismail HI, Chotpitayasunondh T, Chua MN, Luong CQ, Rusmil K, Wirawan DN, Nallusamy R, Pitisuttithum P, Thisyakorn U, Yoon IK, van der Vliet D, Langevin E, Laot T, Hutagalung Y, Frago C, Boaz M, Wartel TA, Tornieporth NG, Saville M, Bouckenooghe A; CYD14 Study Group. Clinical efficacy and safety of a novel tetravalent dengue vaccine in healthy children in Asia: a phase 3, randomised, observer-masked, placebo-controlled trial. Lancet. 2014 Oct 11;384(9951):1358-65. doi: 10.1016/S0140-6736(14)61060-6. Epub 2014 Jul 10. PMID 25018116
- [Background] Villar L, Dayan GH, Arredondo-Garcia JL, Rivera DM, Cunha R, Deseda C, Reynales H, Costa MS, Morales-Ramirez JO, Carrasquilla G, Rey LC, Dietze R, Luz K, Rivas E, Miranda Montoya MC, Cortes Supelano M, Zambrano B, Langevin E, Boaz M, Tornieporth N, Saville M, Noriega F; CYD15 Study Group. Efficacy of a tetravalent dengue vaccine in children in Latin America. N Engl J Med. 2015 Jan 8;372(2):113-23. doi: 10.1056/NEJMoa1411037. Epub 2014 Nov 3. PMID 25365753
- [Background] Guy B, Lang J, Saville M, Jackson N. Vaccination Against Dengue: Challenges and Current Developments. Annu Rev Med. 2016;67:387-404. doi: 10.1146/annurev-med-091014-090848. Epub 2015 Oct 23. PMID 26515983
- [Background] Hadinegoro SR, Arredondo-Garcia JL, Capeding MR, Deseda C, Chotpitayasunondh T, Dietze R, Muhammad Ismail HI, Reynales H, Limkittikul K, Rivera-Medina DM, Tran HN, Bouckenooghe A, Chansinghakul D, Cortes M, Fanouillere K, Forrat R, Frago C, Gailhardou S, Jackson N, Noriega F, Plennevaux E, Wartel TA, Zambrano B, Saville M; CYD-TDV Dengue Vaccine Working Group. Efficacy and Long-Term Safety of a Dengue Vaccine in Regions of Endemic Disease. N Engl J Med. 2015 Sep 24;373(13):1195-206. doi: 10.1056/NEJMoa1506223. Epub 2015 Jul 27. PMID 26214039
- [Background] Schilte C, Staikowsky F, Couderc T, Madec Y, Carpentier F, Kassab S, Albert ML, Lecuit M, Michault A. Chikungunya virus-associated long-term arthralgia: a 36-month prospective longitudinal study. PLoS Negl Trop Dis. 2013;7(3):e2137. doi: 10.1371/journal.pntd.0002137. Epub 2013 Mar 21. PMID 23556021
- [Background] Rolph MS, Foo SS, Mahalingam S. Emergent chikungunya virus and arthritis in the Americas. Lancet Infect Dis. 2015 Sep;15(9):1007-1008. doi: 10.1016/S1473-3099(15)00231-5. No abstract available. PMID 26333330
- [Background] Weaver SC, Costa F, Garcia-Blanco MA, Ko AI, Ribeiro GS, Saade G, Shi PY, Vasilakis N. Zika virus: History, emergence, biology, and prospects for control. Antiviral Res. 2016 Jun;130:69-80. doi: 10.1016/j.antiviral.2016.03.010. Epub 2016 Mar 18. PMID 26996139
- [Background] World Health Organization. WHO Director-General summarizes the outcome of the Emergency Committee regarding clusters of microcephaly and Guillain-Barré syndrome. 2016. Available at. see World Health Organization. Zika virus: Fact sheet. 2016.
- [Background] World Health Organization. Mosquito (vector) control emergency response and preparedness for Zika virus. (2016). Available at: http://www.who.int/neglected_diseases/news/mosquito_vector_control_response/en/. (Accessed: 18th March 2016)
- [Background] Republic of Colombia, B. of the R. (Bogotá). D. of E. R. Colombia: Overview of its economic structure. (Printing of the Bank of the Republic, 1992).
- [Background] Republic of Colombia, N. C. for E. and S. P. Guidelines for the formulation of integral environmental health policy with emphasis on the components of air quality, water quality and chemical safety. (2008).
- [Background] Medina ÁM. El Dengue en Colombia. Epidemiología de la Reemergencia a la Hiperendemia. Medicina. 2013 Mar 5;35(1):75-6.n Ltda. Bogotá).
- [Background] National Institute of Health. Epidemiological bulletin: week 52/2016. (2016).
- [Background] Bowman LR, Donegan S, McCall PJ. Is Dengue Vector Control Deficient in Effectiveness or Evidence?: Systematic Review and Meta-analysis. PLoS Negl Trop Dis. 2016 Mar 17;10(3):e0004551. doi: 10.1371/journal.pntd.0004551. eCollection 2016 Mar. PMID 26986468
- [Background] Andersson N, Nava-Aguilera E, Arostegui J, Morales-Perez A, Suazo-Laguna H, Legorreta-Soberanis J, Hernandez-Alvarez C, Fernandez-Salas I, Paredes-Solis S, Balmaseda A, Cortes-Guzman AJ, Serrano de Los Santos R, Coloma J, Ledogar RJ, Harris E. Evidence based community mobilization for dengue prevention in Nicaragua and Mexico (Camino Verde, the Green Way): cluster randomized controlled trial. BMJ. 2015 Jul 8;351:h3267. doi: 10.1136/bmj.h3267. PMID 26156323
- [Background] Degener CM, Eiras AE, Azara TM, Roque RA, Rosner S, Codeco CT, Nobre AA, Rocha ES, Kroon EG, Ohly JJ, Geier M. Evaluation of the effectiveness of mass trapping with BG-sentinel traps for dengue vector control: a cluster randomized controlled trial in Manaus, Brazil. J Med Entomol. 2014 Mar;51(2):408-20. doi: 10.1603/me13107. PMID 24724291
- [Background] Wilson AL, Boelaert M, Kleinschmidt I, Pinder M, Scott TW, Tusting LS, Lindsay SW. Evidence-based vector control? Improving the quality of vector control trials. Trends Parasitol. 2015 Aug;31(8):380-90. doi: 10.1016/j.pt.2015.04.015. Epub 2015 May 19. PMID 25999026
- [Background] O'Neill SL, Pettigrew MM, Sinkins SP, Braig HR, Andreadis TG, Tesh RB. In vitro cultivation of Wolbachia pipientis in an Aedes albopictus cell line. Insect Mol Biol. 1997 Feb;6(1):33-9. doi: 10.1046/j.1365-2583.1997.00157.x. PMID 9013253
- [Background] Stouthamer R, Breeuwer JA, Hurst GD. Wolbachia pipientis: microbial manipulator of arthropod reproduction. Annu Rev Microbiol. 1999;53:71-102. doi: 10.1146/annurev.micro.53.1.71. PMID 10547686
- [Background] Rousset F, Vautrin D, Solignac M. Molecular identification of Wolbachia, the agent of cytoplasmic incompatibility in Drosophila simulans, and variability in relation with host mitochondrial types. Proc Biol Sci. 1992 Mar 23;247(1320):163-8. doi: 10.1098/rspb.1992.0023. PMID 1350096
- [Background] Hilgenboecker K, Hammerstein P, Schlattmann P, Telschow A, Werren JH. How many species are infected with Wolbachia?--A statistical analysis of current data. FEMS Microbiol Lett. 2008 Apr;281(2):215-20. doi: 10.1111/j.1574-6968.2008.01110.x. Epub 2008 Feb 28. PMID 18312577
- [Background] McMeniman CJ, Lane RV, Cass BN, Fong AW, Sidhu M, Wang YF, O'Neill SL. Stable introduction of a life-shortening Wolbachia infection into the mosquito Aedes aegypti. Science. 2009 Jan 2;323(5910):141-4. doi: 10.1126/science.1165326. PMID 19119237
- [Background] Joubert DA, Walker T, Carrington LB, De Bruyne JT, Kien DH, Hoang Nle T, Chau NV, Iturbe-Ormaetxe I, Simmons CP, O'Neill SL. Establishment of a Wolbachia Superinfection in Aedes aegypti Mosquitoes as a Potential Approach for Future Resistance Management. PLoS Pathog. 2016 Feb 18;12(2):e1005434. doi: 10.1371/journal.ppat.1005434. eCollection 2016 Feb. PMID 26891349
- [Background] Walker T, Johnson PH, Moreira LA, Iturbe-Ormaetxe I, Frentiu FD, McMeniman CJ, Leong YS, Dong Y, Axford J, Kriesner P, Lloyd AL, Ritchie SA, O'Neill SL, Hoffmann AA. The wMel Wolbachia strain blocks dengue and invades caged Aedes aegypti populations. Nature. 2011 Aug 24;476(7361):450-3. doi: 10.1038/nature10355. PMID 21866159
- [Background] Dutra HL, Rocha MN, Dias FB, Mansur SB, Caragata EP, Moreira LA. Wolbachia Blocks Currently Circulating Zika Virus Isolates in Brazilian Aedes aegypti Mosquitoes. Cell Host Microbe. 2016 Jun 8;19(6):771-4. doi: 10.1016/j.chom.2016.04.021. Epub 2016 May 4. PMID 27156023
- [Background] Johnson KN. The Impact of Wolbachia on Virus Infection in Mosquitoes. Viruses. 2015 Nov 4;7(11):5705-17. doi: 10.3390/v7112903. PMID 26556361
- [Background] Rainey SM, Shah P, Kohl A, Dietrich I. Understanding the Wolbachia-mediated inhibition of arboviruses in mosquitoes: progress and challenges. J Gen Virol. 2014 Mar;95(Pt 3):517-530. doi: 10.1099/vir.0.057422-0. Epub 2013 Dec 16. PMID 24343914
- [Background] Amuzu HE, Simmons CP, McGraw EA. Effect of repeat human blood feeding on Wolbachia density and dengue virus infection in Aedes aegypti. Parasit Vectors. 2015 Apr 24;8:246. doi: 10.1186/s13071-015-0853-y. PMID 25903749
- [Background] Ye YH, Carrasco AM, Frentiu FD, Chenoweth SF, Beebe NW, van den Hurk AF, Simmons CP, O'Neill SL, McGraw EA. Wolbachia Reduces the Transmission Potential of Dengue-Infected Aedes aegypti. PLoS Negl Trop Dis. 2015 Jun 26;9(6):e0003894. doi: 10.1371/journal.pntd.0003894. eCollection 2015. PMID 26115104
- [Background] Frentiu FD, Zakir T, Walker T, Popovici J, Pyke AT, van den Hurk A, McGraw EA, O'Neill SL. Limited dengue virus replication in field-collected Aedes aegypti mosquitoes infected with Wolbachia. PLoS Negl Trop Dis. 2014 Feb 20;8(2):e2688. doi: 10.1371/journal.pntd.0002688. eCollection 2014 Feb. PMID 24587459
- [Background] Moreira LA, Iturbe-Ormaetxe I, Jeffery JA, Lu G, Pyke AT, Hedges LM, Rocha BC, Hall-Mendelin S, Day A, Riegler M, Hugo LE, Johnson KN, Kay BH, McGraw EA, van den Hurk AF, Ryan PA, O'Neill SL. A Wolbachia symbiont in Aedes aegypti limits infection with dengue, Chikungunya, and Plasmodium. Cell. 2009 Dec 24;139(7):1268-78. doi: 10.1016/j.cell.2009.11.042. PMID 20064373
- [Background] Ferguson NM, Kien DT, Clapham H, Aguas R, Trung VT, Chau TN, Popovici J, Ryan PA, O'Neill SL, McGraw EA, Long VT, Dui le T, Nguyen HL, Chau NV, Wills B, Simmons CP. Modeling the impact on virus transmission of Wolbachia-mediated blocking of dengue virus infection of Aedes aegypti. Sci Transl Med. 2015 Mar 18;7(279):279ra37. doi: 10.1126/scitranslmed.3010370. PMID 25787763
- [Background] Lessler J, Salje H, Grabowski MK, Cummings DA. Measuring Spatial Dependence for Infectious Disease Epidemiology. PLoS One. 2016 May 19;11(5):e0155249. doi: 10.1371/journal.pone.0155249. eCollection 2016. PMID 27196422
- [Background] Dengue: Guidelines for Diagnosis, Treatment, Prevention and Control: New Edition. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK143157/ PMID 23762963
- [Derived] Velez ID, Tanamas SK, Arbelaez MP, Kutcher SC, Duque SL, Uribe A, Zuluaga L, Martinez L, Patino AC, Barajas J, Munoz E, Mejia Torres MC, Uribe S, Porras S, Almanza R, Pulido H, O'Neill SL, Santacruz-Sanmartin E, Gonzalez S, Ryan PA, Denton JA, Jewell NP, Dufault SM, Simmons CP, Anders KL. Reduced dengue incidence following city-wide wMel Wolbachia mosquito releases throughout three Colombian cities: Interrupted time series analysis and a prospective case-control study. PLoS Negl Trop Dis. 2023 Nov 30;17(11):e0011713. doi: 10.1371/journal.pntd.0011713. eCollection 2023 Nov. PMID 38032857
- [Derived] Velez ID, Santacruz E, Kutcher SC, Duque SL, Uribe A, Barajas J, Gonzalez S, Patino AC, Zuluaga L, Martinez L, Munoz E, Mejia MC, Arbelaez MP, Pulido H, Jewell NP, Dufault SM, O'Neill SL, Simmons CP, Anders KL, Tanamas SK. The impact of city-wide deployment of Wolbachia-carrying mosquitoes on arboviral disease incidence in Medellin and Bello, Colombia: study protocol for an interrupted time-series analysis and a test-negative design study. F1000Res. 2019 Aug 1;8:1327. doi: 10.12688/f1000research.19858.2. eCollection 2019. PMID 34900237
- See also: PECET Web Page — http://pecet-colombia.org/

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03631719/SAP_000.pdf